CLINICAL TRIAL: NCT05897320
Title: Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Intravenous (IV) Eptinezumab in Paediatric Patients (6 to 17 Years) for the Preventive Treatment of Episodic Migraine
Brief Title: A Study of Eptinezumab in Pediatric Participants With Episodic Migraine
Acronym: PROSPECT-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19357A; 2022-502538-14-00 (Other: EU CTR)
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Episodic Migraine
MeSH Terms: interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Eptinezumab 300 mg (Experimental): Participants will receive a single intravenous (IV) infusion of eptinezumab 300 mg (weight adjusted).
  Interventions: Drug: Eptinezumab
- Placebo (Placebo Comparator): Participants will receive a single IV infusion of matching placebo to eptinezumab.
  Interventions: Drug: Placebo
- Eptinezumab 100 mg (Experimental): Participants will receive a single IV infusion of eptinezumab 100 mg (weight adjusted).
  Interventions: Drug: Eptinezumab

INTERVENTIONS:
Drug: Eptinezumab — Solution for infusion
  Arms: Eptinezumab 100 mg; Eptinezumab 300 mg
Drug: Placebo — Solution for infusion
  Arms: Placebo

SUMMARY:
The main goal of this trial is to learn whether eptinezumab helps reduce the number of days with episodic migraine in pediatric participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine (with or without aura) according to the International Classification of Headache Disorders, 3rd edition (ICHD-3; in the opinion of the investigator) with history of migraine headaches of at least 6 months prior to the Screening Visit.
* During the 28-day screening period, the participant (and their parent/caregiver, when applicable) must adequately complete the headache eDiary (≥23 of the 28 days) following the day of the Screening Visit.
* During the 28-day screening period, the participant must have ≤14 headache days, of which at least 4 are migraine days as documented in the eDiary.

Exclusion Criteria:

* History or diagnosis of chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or unusual migraine subtypes (previously referred to as complicated migraine), such as hemiplegic migraine (sporadic and familial), migraine with brainstem aura, recurrent painful ophthalmic neuropathy, or migraine with neurological accompaniments that are not typical of migraine aura (diplopia, altered consciousness, or long duration, e.g., >60 min).
* History of moderate or severe head trauma or other neurological disorder or systemic medical disease that is, in the investigator's opinion, likely to affect the functions of the central nervous system.
* Current psychiatric condition that is uncontrolled and/or untreated for a minimum of 6 months prior to the Screening Visit. Participants with a lifetime history of psychosis and/or mania are excluded.
* Any other disorder for which the treatment takes priority over treatment of migraine or is likely to interfere with study treatment or impair treatment compliance.

Other inclusion and exclusion criteria may apply.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 315 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2027-07-06 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Number of Monthly Migraine Days (MMDs) Averaged Over Weeks 1-12 | Baseline, Weeks 1-12

SECONDARY OUTCOMES:
Response: ≥50% Reduction From Baseline in MMDs | Baseline, Weeks 1-4 and Weeks 1-12
Percentage of Participants with Migraine on the Day After Dosing (Day 1) | On Day After Dosing
Change From Baseline in MMDs with Acute Medication Use | Baseline, Weeks 1-12
Response: ≥75% reduction from baseline in MMDs | Baseline, Weeks 1-4 and Weeks 1-12
Change From Baseline in the Number of Monthly Headache Days (MHDs) | Baseline, Weeks 1-12
Change From Baseline in Monthly Hours with Headache | Baseline, Weeks 1-12
Change From Baseline in Days with Acute Medication | Baseline, Weeks 1-12
Change From Baseline in Rate of Migraines with Severe Pain Intensity | Baseline, Weeks 1-12
Change From Baseline to Week 12 in Pediatric Migraine Disability Assessment (PedMIDAS) Score | Baseline, Week 12
Free Eptinezumab Plasma Concentrations | Day 0 (pre-dose) and at Weeks 8, 12, and 20
Number of Participants With Specific Anti-eptinezumab Antibodies (Anti-Drug Antibodies [ADA]) | Day 0 (pre-dose) and at Weeks 8, 12, and 20
Number of Participants With Specific ADA-Positive Samples for Neutralizing Antibodies (NAb) | Day 0 (pre-dose) and at Weeks 8, 12, and 20

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — HQ_Medinfo@Lundbeck.com
Locations (63):
- United States (14):
  - Ki Health Partners LLC DBA New England Institute for Clinical Research, Stamford, Connecticut
  - Child Neurology of NW Florida, Gulf Breeze, Florida
  - A G A Clinical Trials, Hialeah, Florida
  - University of South Florida, Tampa, Florida
  - University of Kentucky HealthCare (UKHC) Kentucky Clinic, Lexington, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - North Suffolk Neurology-Commack, Commack, New York
  - OnSite Clinical Solutions, LLC - Randolph Rd - Charlotte, Charlotte, North Carolina
  - Childrens Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center - PIN, Cincinnati, Ohio
  - Road Runner Research Ltd, San Antonio, Texas
  - Children's Specialty Group - 3 Commercial Place, Norfolk, Virginia
  - Childrens Hospital of Wisconsin - PIN, New Berlin, Wisconsin
- Argentina (7):
  - Clínica Privada Independencia, Munro, Buenos Aires
  - Hospital Britanico de Buenos Aires, Barracas, Ciudad Autónoma de BuenosAires
  - Expertia S.A- Mautalén Salud e Investigación, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - Centro de Investigaciones Médicas Tucumán - PPDS, San Miguel de Tucumán, Tucumán Province
  - Hospital de Niños de La Santisima Trinidad, Córdoba
- Canada (4):
  - Medical Arts Health Research Group - Penticton, Penticton, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - The Kids Clinic, Ajax, Ontario
  - London Health Sciences Centre -800 Commissioners Rd E, London, Ontario
- Italy (8):
  - Ospedale Pediatrico Bambino Gesù IRCCS, Rome, Lazio
  - Istituto G Gaslini Ospedale Pediatrico IRCCS, Genoa, Liguria
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino IRCCS, Pavia, Lombardy
  - AO Brotzu - Clinica di Neuropsichiatria dell'Infanzia e dell'Adolescenza - INCIPIT - PIN, Cagliari, Sardinia
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa, Tuscany
- Clinical Research Institute SC-Mexico, Tepetlacolco, Mexico
- Poland (7):
  - AthleticoMed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - ETG Neuroscience - PPDS, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Plejady Magdalena Celinska - Lowenhoff, Michal Zolnowski Spolka komandytowa, Krakow
  - ETG Lublin - PPDS, Lublin
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. Sp. k., Oświęcim
  - MTZ Clinical Research Powered by PRATIA - PPDS, Warsaw
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw
- Portugal (5):
  - ULS de Santo António, EPE - Centro Materno Infantil Norte, Porto Covo, Setúbal District
  - Centro Clínico Académico, Braga - Hospital de Braga, Braga
  - ULS de Coimbra, EPE - Hospital Pediátrico de Coimbra, Coimbra
  - Hospital CUF Descobertas, Lisbon
  - ULS de São João, EPE - Hospital de São João, Porto Covo
- Serbia (5):
  - Childrens University Hospital, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
  - Children and Youth Health Care Institute of Vojvodina, Novi Sad
  - Clinical Centre of Vojvodina, Novi Sad
- Spain (4):
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Turkey (Türkiye) (4):
  - Izmir City Hospital, Bayraklı, İzmir
  - Eskisehir Osmangazi Universitesi Tip Fakultesi Hastanesi, Eskişehir
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Fatih/Istanbul
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin
- United Kingdom (4):
  - Royal Hospital for Children (Glasgow) - PPDS - PIN, Glasgow, Glasgow City
  - Royal Hospital for Children and Young People - PIN, Edinburgh, Midlothian
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth, Norfolk
  - Great Ormond Street Hospital, London